CLINICAL TRIAL: NCT04387383
Title: Acupuncture for Irritable Bowel Syndrome Patients: A Single-blinded Randomized Sham-controlled Clinical Trial
Brief Title: Acupuncture for Irritable Bowel Syndrome Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Zhong Lidan, Assistant Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKBU AcupIBS
Record Dates: First submitted 2020-05-03; First posted 2020-05-13 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: single-blinded, randomized, sham-controlled clinical trial
Who Masked: Participant
Masking Description: Subjects of both groups will be randomly assigned to receive either electro-acupuncture or control (sham) treatment. For randomization, simple, complete non-sequential random numbers will be generated in advance by a computer program in a block of four, and kept by the principal investigator. After a patient's eligibility is confirmed, a randomization number which corresponds to the group allocation will be provided to the acupuncturist by the PI. This arrangement will ensure that the clinical assessor and participants are blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture group (Experimental): Electro-acupuncture will be conducted for 2 sessions per week over 6 consecutive weeks. Disposable acupuncture needles (0.30 mm in diameter and 25-40 mm in length) are inserted at a depth of 10-30 mm obliquely into scalp acupuncture points (Baihui, Toulinqi) or straightly into body acupuncture points (Taichong, Zhangmen, Sanyinjiao, Zhongwan, Guanyuan, Tianshu, Zusanli). Electroacupuncture will be applied to the abdominal points at fast and dispersed waves through electric needle stimulator (ES-160 6-Channel Programmable Electro-acupuncture) for 30 min. The intensity is adjusted to a level at which patients feel comfortable.
  Interventions: Device: Acupuncture
- sham-acupuncture group (Placebo Comparator): Sham-acupuncture will be conducted for 2 sessions per week over 6 consecutive weeks. Disposable acupuncture needles (0.30 mm in diameter and 25-40 mm in length) are inserted at the same way as in the acupuncture group but on sham-acupuncture points (Sham-Baihui, Sham-Toulinqi, Sham-Taichong, Sham-Zhangmen, Sham-Sanyinjiao, Sham-Zhongwan, Sham-Guanyuan, Sham-Tianshu, Sham-Zusanli). The sham points are non-acupuncture points nor located on meridians
  Interventions: Device: Sham-acupuncture

INTERVENTIONS:
Device: Acupuncture — Disposable acupuncture needles (0.30 mm in diameter and 25-40 mm in length) are inserted at a depth of 10-30 mm obliquely into scalp acupuncture points (Baihui, Toulinqi) or straightly into body acupuncture points (Taichong, Zhangmen, Sanyinjiao, Zhongwan, Guanyuan, Tianshu, Zusanli). Electroacupuncture will be applied to the abdominal points at fast and dispersed waves through electric needle stimulator (ES-160 6-Channel Programmable Electro-acupuncture) for 30 min. The intensity is adjusted to a level at which patients feel comfortable.
  Arms: Acupuncture group
Device: Sham-acupuncture — Disposable acupuncture needles (0.30 mm in diameter and 25-40 mm in length) are inserted at the same way as in the acupuncture group but on sham-acupuncture points (Sham-Baihui, Sham-Toulinqi, Sham-Taichong, Sham-Zhangmen, Sham-Sanyinjiao, Sham-Zhongwan, Sham-Guanyuan, Sham-Tianshu, Sham-Zusanli). The sham points are non-acupuncture points nor located on meridians
  Arms: sham-acupuncture group

SUMMARY:
In this study, a 14-week, single blinded, randomized controlled clinical trial will be conducted to determine whether acupuncture could have significant benefits than sham acupuncture for IBS.

DETAILED DESCRIPTION:
This is a single blinded randomized sham controlled clinical trial with two arms. 120 IBS patients will be recruited. The study will cooperate with Hong Kong Baptist University, and University of Toronto. After a 2-week run-in period, eligible subjects will be randomly assigned to one of two arms, acupuncture (AC) arm and sham acupuncture (SAC) arm. Each eligible subject will go through a 2-wk run-in-period, 6-wk treatment period and follow by a 6-wk of follow-up period. Five visits in total were scheduled for each subject in week 0, week 2, week 5, week 8 and week 14.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of the Rome IV criteria for IBS
* IBS Symptom Severity Scale (IBS-SSS) > 75 points (a range of 0-500 points of VAS on five questions) at baseline and during the 2-week run-in period
* Written informed consent.

Exclusion Criteria:

* Pregnancy or breast-feeding
* Medical history of inflammatory bowel diseases, carbohydrate malabsorption, hormonal disorder, known allergies to food additives, and/or any other serious diseases
* Unstable medical conditions
* Unstable mental condition or with history of mental illness
* Patients who have received acupuncture treatment in last three months, or took concomitant medication with affect gastrointestinal motility or visceral sensation, such as antidiarrheal agent, antidepressant, narcotic analgesic, and anticholinergic
* Alcoholism or drug abuse in past 1 year
* Having needle phobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change on IBS-symptom severity scale | 0,8,14 weeks
  Value from 0-500. The higher the score, the more severe the symptoms. When there is lowering of the sore between baseline and treatments, it indicates clinical improvement.
Change on Hamilton Depression Rating Scale (HAMD-17) | 0,8,14 weeks
  Value from 0-57. Scoring 8-16: mild depression, 17-23: moderate depression, over 24: severe depression. When there is lowering of the sore between baseline and treatments, it indicates improvement on depressive symptoms.
Change on Clinical Global Impression-severity (CGI-S) | 0,8,14 weeks
  Rating from 1-7, the higher rate indicates more severe of the mental problem. The subject is rated by researcher from his clinical experience. When there is lowering of the rating between baseline and treatments, it indicates improvement.
Change on Self-Rating Depression Scale (SDS) | 0,8,14 weeks
  Value from 20-80. Scoring 50-69: depression, over 70: severe depression. When there is lowering of the sore between baseline and treatments, it indicates improvement.
Change on IBS Quality of Life (IBS-QoL) | 0,8,14 weeks
  Value from 35-170. The higher the score, the lower the quality of life. When there is lowering of the sore between baseline and treatments, it indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoxiang Bian, MD., Ph.D, Study Director — Hong Kong Chinese Medicine Clinical Study Centre
Locations (1):
- Linda Zhong, Kowloon Tong, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhong LLD, Lam TF, Yang W, Zheng Y, Lyu Z, Bian Z. Electro-acupuncture for irritable bowel syndrome patients: study protocol for a single-blinded randomized sham-controlled clinical trial. Trials. 2021 Sep 15;22(1):619. doi: 10.1186/s13063-021-05563-4. PMID 34526079